CLINICAL TRIAL: NCT01798017
Title: Introducing Mifepristone-Misoprostol for Menstrual Regulation in Public Sector Facilities in Bangladesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1004
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2013-03

CONDITIONS: Menstrual Regulation
Keywords: menstrual regulation; mifepristone; misoprostol
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mifepristone-misoprostol (Experimental): Women will receive 200mg oral mifepristone followed in 24-48h by 800mcg buccal misoprostol
  Interventions: Drug: Mifepristone and misoprostol

INTERVENTIONS:
Drug: Mifepristone and misoprostol — Women will receive 200mg mifepristone followed in 24-48h by 800mcg bucccal misoprsotol

SUMMARY:
This open-label study is being conducted to determine whether a mifepristone-misoprostol regimen for uterine evacuation which consists of 200 mg mifepristone followed 24 hours later by 800 mcg buccal misoprostol is acceptable to women and providers and feasible for introduction in public sector facilities in Bangladesh. It will also determine the feasibility of women availing the option of taking their dose of misoprostol outside the facility.

DETAILED DESCRIPTION:
This open-label study is being conducted to determine whether a mifepristone-misoprostol regimen for uterine evacuation which consists of 200 mg mifepristone followed 24 hours later by 800 mcg buccal misoprostol is acceptable to women and providers and feasible for introduction in public sector facilities in Bangladesh. It will also determine the feasibility of women availing the option of taking their dose of misoprostol outside the facility.

The specific aims of this project are as follows:

* Assess whether a uterine evacuation regimen that allows women the option of taking their misoprostol outside the facility and which consists of 200 mg mifepristone followed 24 hours later by 800 mcg buccal misoprostol is feasible for introduction in a range of clinical settings in government facilities in Bangladesh;
* Determine whether a mifepristone-misoprostol regimen for uterine evacuation is acceptable to women and providers; and
* Determine what proportion of women, if offered the choice, would prefer to take misoprostol in the facility and what proportion would prefer to take it outside the facility.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to sign consent forms;
* Be eligible for menstrual regulation (MR) services according to clinician's assessment;
* Be willing to undergo a surgical evacuation if necessary;
* Be willing to provide a urine sample prior to administration of the mifepristone
* Have ready and easy access to a telephone and
* Agree to comply with the study procedures and visit schedule

Exclusion Criteria:

* • Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass;

  * Chronic renal failure;
  * Concurrent long-term corticosteroid therapy;
  * History of allergy to mifepristone, misoprostol or other prostaglandin;
  * Hemorrhagic disorders or concurrent anticoagulant therapy;
  * Inherited porphyrias; or
  * Other serious physical or mental health conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1738 (Actual)
Dates: Start 2012-11; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
successful menstrual regulation without the need for a surgical evacuation | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Hillary J Bracken, PhD, Principal Investigator — Gynuity Health Projects; Laura Reichenbach, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (8):
- Bangladesh (8):
  - Aminbazar Rural Dispensary, Aminbazar, Dhaka Division
  - MCH-Unit, Upazilla Health Center, Savar Upazila, Dhaka Division
  - Tetulzhora UH&FWC, Tetuljhora, Dhaka Division
  - Chartarapur UH & FWC, Chandrapur, Rajshahi Division
  - Goyeshpur UH &FWC, Goyespur, Rajshahi Division
  - MCH Unit, Sadar Upazilla, Pābna, Rajshahi Division
  - Pabna MCWC, Pābna, Rajshahi Division
  - Mohammadpur Fertility Services and Training Center, Dhaka

REFERENCES:
- [Derived] Alam A, Lotarevich T, Das TR, Reichenbach L, Bracken H. Mifepristone-misoprostol for menstrual regulation in public sector facilities in Bangladesh. Int J Gynaecol Obstet. 2018 Feb;140(2):205-210. doi: 10.1002/ijgo.12356. Epub 2017 Nov 9. PMID 29049861